CLINICAL TRIAL: NCT04240457
Title: Safety and Effectiveness of the PXL-Platinum 330 System for Corneal Crosslinking in Eyes With Corneal Ectatic Conditions
Brief Title: Safety and Efficacy of Corneal Crosslinking Using the PXL-Platinum 330 for Eyes With Corneal Ectatic Conditions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to enrollment and other challenges attributable to the Covid-19 public health emergency.
Sponsor: Arbor Center for Eye Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 330019
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Keratoconus; Cornea Ectasia
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: Treatment of patients with disease
Who Masked: Outcomes Assessor
Masking Description: Randomized at outset
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Pulsed, accelerated (Experimental): 18mW, 5 seconds on, 5 seconds off, 10 minutes of illumination.
  Interventions: Combination Product: Epithelial-on Corneal Crosslinking with the PXL 330 Platinum system.
- Conventional (Active Comparator): 9mW continuous, 10 minutes of illumination.
  Interventions: Combination Product: Epithelial-on Corneal Crosslinking with the PXL 330 Platinum system.

INTERVENTIONS:
Combination Product: Epithelial-on Corneal Crosslinking with the PXL 330 Platinum system. — PXL-330 Platinum device for crosslinking with Peschke riboflavin solution. Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea.

SUMMARY:
To evaluate the safety and effectiveness of the PXL Platinum 330 device for performing Corneal Crosslinking in patients with corneal thinning conditions.

DETAILED DESCRIPTION:
Patients with progressive keratoconus, pellucid marginal degeneration, or at risk for post-refractive corneal ectasia will be recruited and undergo epithelial-on corneal crosslinking with the Peschke PXL-330 system using pulsed, accelerated energy delivery. Patients will undergo monitoring for 1 year, with serial measurements of corneal topography, visual acuity, intraocular pressure and visual function questionnaire assessments.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: Criterion 1,2,3 are required for all participants. Participants must also meet one or more of criteria 4-12 . Criterion 13 is relevant only for contact lens wearers

Subjects who have one or both eyes that meet criteria 1 and one or more of the following criteria will be considered candidates for this study:

1. 12 years of age or older
2. Presence of central or inferior steepening.
3. Axial topography consistent with keratoconus, post-surgical ectasia, or pellucid marginal degeneration
4. Presence of one or more findings associated with keratoconus or pellucid marginal degeneration, such as:

   1. Fleischer ring
   2. Vogt's striae
   3. Decentered corneal apex
   4. Munson's sign
   5. Rizzutti's sign
   6. Apical Corneal scarring consistent with Bowman's breaks
   7. Scissoring of the retinoscopic reflex
   8. Crab-claw appearance on topography
5. Steepest keratometry (Kmax) value ≥ 47.20 D
6. I-S keratometry difference > 1.5 D on the Pentacam map
7. Posterior corneal elevation >16 microns
8. Thinnest corneal point <485 microns
9. Predicted Post LASIK/PRK stromal ablation depth <350 microns or expected keratometry >47.2 D, or patients undergoing PRK in keratoconus suspect eyes
10. Contact Lens Wearers Only:

    a. Removal of contact lenses for the required period of time prior to the screening refraction:
11. Signed written informed consent
12. Willingness and ability to comply with schedule for follow-up visits
13. Contact Lens Wearers Only:

    1. Removal of contact lenses for the required period of time prior to the screening refraction:

Contact Lens Type Minimum Discontinuation Time: Soft 1 Week, Soft Extended Wear 2 Weeks, Soft Toric 3 Weeks, Rigid Gas Permeable 2 Weeks per decade of wear

Exclusion Criteria (any of the following are reasons for exclusion):

1. Eyes classified as either normal or atypical normal on the severity grading scheme.
2. Corneal pachymetry at the screening exam that is <300 microns at the thinnest point in the eye(s) to be treated.
3. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example:

   1. History of or active corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, acanthamoeba, etc.)
   2. Clinically significant corneal scarring in the CXL treatment zone that is not related to keratoconus, or in the investigator's opinion, will interfere with the cross-linking procedure.
4. Pregnancy (including plan to become pregnant) or lactation during the course of the study
5. A known sensitivity to study medications
6. Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests.
7. Patients with a current condition that, in the physician's opinion, would interfere with or prolong epithelial healing

   -

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2023-02-18 (Actual); Study Completion 2023-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lubeck, MD, Principal Investigator — Arbor Center for Eye Care
Locations (1):
- Arbor Center for Eye Care, Orland Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Groups:
- Pulsed, Accelerated: 18mW, 5 seconds on, 5 seconds off, 10 minutes of illumination.
  Epithelial-on Corneal Crosslinking with the PXL 330 Platinum system.: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution.
  Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea.
- Conventional: 9mW continuous, 10 minutes of illumination.
  Epithelial-on Corneal Crosslinking with the PXL 330 Platinum system.: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution.
  Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea.
Period: Overall Study
Arm/Group | Pulsed, Accelerated | Conventional
Started | 7; 13 Eyes | 4; 4 Eyes
Completed | 2; 4 Eyes | 3; 3 Eyes
Not Completed | 5; 9 Eyes | 1; 1 Eyes
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Population: Patients recruited at a single center based on physician examination for corneal ectasia in one or both eyes. The first patient was screened for enrollment in June 2020, while the last patient was screened in October 2021.
Units Other Than Participants: Eyes
Groups:
- Pulsed, Accelerated: Following riboflavin instillation, the eye was exposed to UVA pulsed light at 18mW/cm2 for 5 seconds, followed by 5 seconds off, repeating over 10 minutes of illumination.
  Epithelial-on Corneal Crosslinking with the PXL 330 Platinum system.: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution.
  Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea.
- Conventional: Following riboflavin instillation, the eye was exposed to UVA continuous light at 9mW/cm2 for 10 minutes
  Epithelial-on Corneal Crosslinking with the PXL 330 Platinum system.: PXL-330 Platinum device for crosslinking with Peschke riboflavin solution.
  Riboflavin will be used to load the cornea, followed by UV-A crosslinking of the cornea.
- Total: Total of all reporting groups
Arm/Group | Pulsed, Accelerated | Conventional | Total
Number analyzed (Participants) | 7 | 4 | 11
Number analyzed (Eyes) | 13 | 4 | 17
Age, Categorical [Count of Units; unit: Eyes]
  <=18 years | 4 | 0 | 4
  Between 18 and 65 years | 9 | 4 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (11.1) | 36.8 (13.2) | 31.2 (11.6)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 10 | 2 | 12
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Keratometry in Diopters
Description: Average keratometry across the anterior topography of the cornea computed by a validated topographer
Time Frame: 1 year
Population: The study was conducted during the COVID-19 pandemic. Some patients were unable or felt uncomfortable presenting to a physician's office for follow-up measurements. These individuals are marked as "lost to follow up"
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: Eyes
Arm/Group | Pulsed, Accelerated | Conventional
Number analyzed (Participants) | 7 | 4
Number analyzed (Eyes) | 13 | 4
Diopters
  Screening | 51.0 (9.9) | 49.8 (4.8)
  3 months: number analyzed (Participants) | 4 | 4
  3 months: number analyzed (Eyes) | 7 | 4
  3 months | 50.3 (7.8) | 49.0 (5.6)
  6 months: number analyzed (Participants) | 2 | 4
  6 months: number analyzed (Eyes) | 4 | 4
  6 months | 46.6 (.9) | 49.1 (5.5)
  12 months: number analyzed (Participants) | 2 | 4
  12 months: number analyzed (Eyes) | 4 | 4
  12 months | 47.9 (11.3) | 45.8 (4.6)

2. Secondary Outcome: Best Corrected Visual Acuity With Spectacles or Contact Lenses
Description: Measurement of best corrected visual acuity on the validated early-treatment diabetic retinopathy study scale. Snellen chart was used. Values closer to 20/20 indicate better vision.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pulsed, Accelerated | Conventional
Number analyzed (Participants) | 7 | 4
Number analyzed (Eyes) | 13 | 4
Eyes
  Screening: 20/25 or better | 0 | 0
  Screening: 20/30 - 20/50 | 0 | 1
  Screening: 20/60 - 20/200 | 8 | 2
  Screening: Worse than 20/200 | 5 | 1
  1 month post-procedure: number analyzed (Participants) | 4 | 3
  1 month post-procedure: number analyzed (Eyes) | 8 | 3
  1 month post-procedure: 20/25 or better | 0 | 1
  1 month post-procedure: 20/30 - 20/50 | 6 | 1
  1 month post-procedure: 20/60 - 20/200 | 2 | 1
  1 month post-procedure: Worse than 20/200 | 0 | 0
  3 months post- procedure: number analyzed (Participants) | 5 | 3
  3 months post- procedure: number analyzed (Eyes) | 9 | 3
  3 months post- procedure: 20/25 or better | 1 | 1
  3 months post- procedure: 20/30 - 20/50 | 6 | 2
  3 months post- procedure: 20/60 - 20/200 | 1 | 0
  3 months post- procedure: Worse than 20/200 | 1 | 0
  6 months post-procedure: number analyzed (Participants) | 3 | 3
  6 months post-procedure: number analyzed (Eyes) | 6 | 3
  6 months post-procedure: 20/25 or better | 1 | 1
  6 months post-procedure: 20/30 - 20/50 | 5 | 1
  6 months post-procedure: 20/60 - 20/200 | 0 | 1
  6 months post-procedure: Worse than 20/200 | 0 | 0
  12 months post-procedure: number analyzed (Participants) | 2 | 3
  12 months post-procedure: number analyzed (Eyes) | 2 | 3
  12 months post-procedure: 20/25 or better | 1 | 1
  12 months post-procedure: 20/30 - 20/50 | 1 | 1
  12 months post-procedure: 20/60 - 20/200 | 0 | 1
  12 months post-procedure: Worse than 20/200 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pulsed, Accelerated | Conventional
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 1/7 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed, Accelerated (N=7) | Conventional (N=4)
Photophobia (Eye disorders) | 1 (1) | NA — Subject complained of increased photophobia at the 1 week post-procedure visit. Noted resolved at the 1 mo. visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04240457/Prot_SAP_000.pdf